CLINICAL TRIAL: NCT03357523
Title: Evaluation of Peripheral Microcirculation Hemodynamics Following Various Changes Based on Noninvasive Thermography: A Prospective, Randomized, Controlled Trial
Brief Title: Evaluation of Peripheral Microcirculation Hemodynamics Following Various Changes Based on Noninvasive Thermography
Acronym: MRT02
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Afeka, The Tel-Aviv Academic College of Engineering (Other)
Collaborators: Hebrew University of Jerusalem (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 05.04.2017-1-AFK
Record Dates: First submitted 2017-11-20; First posted 2017-11-30 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Microcirculation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red LED (Experimental): Light emitting diodes, 633 nm, 70 mW/cm2, Omnilux new-U (Red LED) (Photomedex, Horsham, PA, USA); RESPeRATE; Heating bag
  Interventions: Device: Omnilux new-U (Red LED); Device: RESPeRATE; Device: Heating bag
- Near Infrared LED (Active Comparator): Light emitting diodes, 830 nm, 55 mW/ cm2, Omnilux new-U (Near infrared LED) (Photomedex, Horsham, PA, USA); RESPeRATE metronome; Heating bag
  Interventions: Device: Omnilux new-U (Near infrared LED); Device: RESPeRATE; Device: Heating bag

INTERVENTIONS:
Device: Omnilux new-U (Red LED) — The left wrist (including area of radial artery) will be illuminated with the Omnilux new-U (Red LED) light source, while the right wrist will not be illuminated
  Arms: Red LED
Device: Omnilux new-U (Near infrared LED) — The left wrist (including area of radial artery) will be illuminated with the Omnilux new-U (Near infrared LED) light source, while the right wrist will not be illuminated
  Arms: Near Infrared LED
Device: RESPeRATE — The subjects will be guided by a digital metronome to breath at 15, 10, and 6 breaths/min for 2 minutes each using the metronome function of the device RESPeRATE (InterCure, Israel) that guides breathing using musical tones played at selectable rhythm
Device: Heating bag — Applying a standard 10X13 [cm] heating bag on the surface of the hand at 43-45 degree Celsius for 10 seconds

SUMMARY:
The objective of the current study is to investigate the hemodynamic changes in the peripheral microcirculation system as a response to various changes, using noninvasive thermography and laser doppler

DETAILED DESCRIPTION:
This study includes a single session per subject. Microvascular and systemic variables will be monitored in response to a number of non-invasive interventions/device that are approved for clinical use and known to elicit microvascular responses. These interventions are applied consecutively, include breathing at different rates, low power visible light in the red-to-near-infrared range, increase in local temperature, and changes in the arm position.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females, between 23 and 45 years of age.
2. Willing to sign informed consent

Exclusion Criteria:

1. Currently smoking
2. Any abnormal skin condition in the area of light irradiation.
3. Pregnant having given birth less than 3 months ago, and/or breastfeeding.
4. Having a history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treated area, unless treatment is conducted following a prophylactic regimen.
5. Having any illness that might affect the vasculature, such as diabetes (type I or II)
6. Suffering from significant concurrent illness, such as cardiac disorders or pertinent neurological disorders.
7. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Capillary blood flow | Up to 1 hour
  Capillary blood flow (red blood cell velocity or flux in 'perfusion units') as measured by laser doppler (Biopac™ System, Inc, USA). This is a continuous measurement (at least 10 Hz sampling rate) from baseline to end of experiment.

SECONDARY OUTCOMES:
Temperature distribution over hands measured by thermography | Up to 1 hour
  Thermographic images will be photographed with a FLIR camera and temperature distribution will be analysed. Photos will be taken every minute from baseline to end of experiment.
Tissue oxygenation (tcPO2) | Up to 1 hour
  Tissue oxygenation (tcPO2) measured by electrodes mounted on both hands (Perimed™ system, Sweden). This is a continuous measurement (at least 10 Hz sampling rate) from baseline to end of experiment.

CONTACTS AND LOCATIONS:
Overall Officials: Zehava Blechman, PhD, Principal Investigator — Afeka Tel Aviv Academic College of Engineering
Locations (1):
- Afeka, Tel-Aviv Academic College of Engineering, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gavish L, Hoffer O, Rabin N, Halak M, Shkilevich S, Shayovitz Y, Weizman G, Haim O, Gavish B, Gertz SD, Ovadia-Blechman Z. Microcirculatory Response to Photobiomodulation-Why Some Respond and Others Do Not: A Randomized Controlled Study. Lasers Surg Med. 2020 Nov;52(9):863-872. doi: 10.1002/lsm.23225. Epub 2020 Feb 17. PMID 32064652